CLINICAL TRIAL: NCT04134936
Title: A Phase Ib, Open-label, Randomized Study to Assess Safety and Preliminary Efficacy of Tafasitamab in Addition to R-CHOP or Tafasitamab Plus Lenalidomide in Addition to R-CHOP in Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma (DLBCL) - First-MIND
Brief Title: Phase Ib Study to Assess Safety and Preliminary Efficacy of Tafasitamab or Tafasitamab Plus Lenalidomide in Addition to R-CHOP in Patients With Newly Diagnosed DLBCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOR208C107
Record Dates: First submitted 2019-10-11; First posted 2019-10-22 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL; CD19; monoclonal antibody; tafasitamab; lenalidomide; MOR208; MOR00208
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Tafasitamab in addition to R-CHOP
  Interventions: Drug: Tafasitamab
- Arm B (Experimental): Tafasitamab plus lenalidomide in addition to R-CHOP
  Interventions: Drug: Tafasitamab plus lenalidomide

INTERVENTIONS:
Drug: Tafasitamab — Six 21-day cycles of tafasitamab (12 mg/kg intravenously, on Day 1, 8 and 15) in addition to R-CHOP
  Arms: Arm A
Drug: Tafasitamab plus lenalidomide — Six 21-day cycles of tafasitamab (12 mg/kg intravenously, on Day 1, 8 and 15) plus lenalidomide (starting dose 25 mg orally, on Day 1-10) in addition to R-CHOP
  Arms: Arm B

SUMMARY:
This is an open-label, randomized, multicentre study to evaluate safety and preliminary efficacy of the human anti-CD19 antibody Tafasitamab in addition to R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone) or Tafasitamab and Lenalidomide in addition to R-CHOP in adult patients with newly diagnosed, previously untreated Diffuse Large B-cell Lymphoma (DLBCL).

ELIGIBILITY:
Major Inclusion Criteria:

1. Age >18 years
2. Histologically confirmed diagnosis of DLBCL, not otherwise specified (NOS)
3. Tumor tissue for retrospective central pathology review and correlative studies must be provided.
4. At least one bidimensionally measurable, PET positive disease site (greatest transverse diameter of ≥1.5 cm, greatest perpendicular diameter of ≥1.0 cm)
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
6. International Prognostic Index (IPI) status of 2 to 5
7. Appropriate candidate for R-CHOP
8. Left ventricular ejection fraction (LVEF) of ≥50% assessed by echocardiography or cardiac multi-gated acquisition (MUGA) scan
9. Adequate hematologic, liver and renal function
10. Females of childbearing potential (FCBP) must:

    * not be pregnant
    * refrain from breast feeding and donating oocyte
    * agree to ongoing pregnancy testing
    * commit to continued abstinence from heterosexual intercourse, or agree to use and be able to comply with the use of double-barrier contraception
11. Males must:

    * use an effective barrier method of contraception if sexually active with FCBP
    * refrain from donating sperm
12. In the opinion of investigator, the patient must be able and willing to receive adequate prophylaxis and/or therapy for thromboembolic events

Major Exclusion Criteria:

1. Any other histological type of lymphoma according to World Health Organization (WHO) 2016 classification of lymphoid neoplasms, known double- or triple-hit lymphoma
2. Transformed non-Hodgkin lymphoma (NHL) and/or evidence of composite lymphoma
3. History of radiation therapy to ≥25% of the bone marrow or history of anthracycline therapy
4. History of prior non-hematologic malignancy except for the following:

   * Malignancy treated with curative intent and with no evidence of active disease present for more than 2 years before screening
   * Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled non-melanomatous skin cancer
   * Adequately treated carcinoma in situ without current evidence of disease
5. History of myocardial infarction ≤6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening arrhythmias
6. Patients with:

   * positive test results for active hepatitis B and C
   * known seropositive for or history of active viral infection with human immunodeficiency virus (HIV)
   * known active bacterial, viral, fungal, mycobacterial, or other infection at screening
   * known central nervous system (CNS) lymphoma involvement
   * history or evidence of clinically significant cardiovascular, CNS and/or other systemic disease that would in the investigator opinion preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (23):
  - MorphoSys Research Site, Tucson, Arizona
  - MorphoSys Research Site, Anaheim, California
  - MorphoSys Research Site, Duarte, California
  - MorphoSys Research Site, Encinitas, California
  - MorphoSys Research Site, Aurora, Colorado
  - MorphoSys Research Site, New Haven, Connecticut
  - MorphoSys Research Site, Washington D.C., District of Columbia
  - MorphoSys Research Site, Urbana, Illinois
  - MorphoSys Research Site, Louisville, Kentucky
  - MorphoSys Research Site, Covington, Louisiana
  - MorphoSys Research Site, Rockville, Maryland
  - MorphoSys Research Site, Ann Arbor, Michigan
  - MorphoSys Research Site, Rochester, Minnesota
  - MorphoSys Research Site, Cincinnati, Ohio
  - MorphoSys Research Site, Cleveland, Ohio
  - MorphoSys Research Site, Eugene, Oregon
  - MorphoSys Research Site, Charleston, South Carolina
  - MorphoSys Research Site, Austin, Texas
  - MorphoSys Research Site, Dallas, Texas
  - MorphoSys Research Site, Houston, Texas
  - MorphoSys Research Site, San Antonio, Texas
  - MorphoSys Research Site, Tyler, Texas
  - MorphoSys Research Site, Vancouver, Washington
- Austria (7):
  - MorphoSys Research Site, Graz
  - MorphoSys Research Site, Innsbruck
  - MorphoSys Research Site, Linz
  - MorphoSys Research Site, Salzburg
  - MorphoSys Research Site, Sankt Pölten
  - MorphoSys Research Site, Vienna
  - MorphoSys Research Site, Wels
- Belgium (5):
  - MorphoSys Research Site, Antwerp
  - MorphoSys Research Site, Brussels
  - MorphoSys Research Site, Ghent
  - MorphoSys Research Site, Roeselare
  - MorphoSys Research Site, Yvoir
- Czechia (3):
  - MorphoSys Research Site, Hradec Králové
  - MorphoSys Research Site, Ostrava
  - MorphoSys Research Site, Prague
- France (4):
  - MorphoSys Research Site, Bordeaux
  - MorphoSys Research Site, Brest
  - MorphoSys Research Site, Nantes
  - MorphoSys Research Site, Pierre-Bénite
- Germany (11):
  - MorphoSys Research Site, Aachen
  - MorphoSys Research Site, Augsburg
  - MorphoSys Research Site, Bonn
  - MorphoSys Research Site, Dortmund
  - MorphoSys Research Site, Giessen
  - MorphoSys Research Site, Göttingen
  - MorphoSys Research Site, Halle
  - MorphoSys Research Site, Mutlangen
  - MorphoSys Research Site, München
  - MorphoSys Research Site, Nuremberg
  - MorphoSys Research Site, Würzburg
- Italy (2):
  - MorphoSys Research Site, Bologna
  - MorphoSys Research Site, Ravenna
- Portugal (2):
  - MorphoSys Research Site, Lisbon
  - MorphoSys Research Site, Porto
- Spain (7):
  - MorphoSys Research Site, Barcelona
  - MorphoSys Research Site, Cáceres
  - MorphoSys Research Site, Girona
  - MorphoSys Research Site, Madrid
  - MorphoSys Research Site, Sabadell
  - MorphoSys Research Site, Seville
  - MorphoSys Research Site, Vitoria-Gasteiz

REFERENCES:
- [Derived] Roschewski M, Kurtz DM, Westin JR, Lynch RC, Gopal AK, Alig SK, Sworder BJ, Cherng HJ, Kuffer C, Blair D, Brown K, Goldstein JS, Schultz A, Close S, Chabon JJ, Diehn M, Wilson WH, Alizadeh AA. Remission Assessment by Circulating Tumor DNA in Large B-Cell Lymphoma. J Clin Oncol. 2025 Dec;43(34):3652-3661. doi: 10.1200/JCO-25-01534. Epub 2025 Aug 13. PMID 40802906
- [Derived] Belada D, Kopeckova K, Bergua Burgues JM, Stevens D, Andre M, Persona EP, Pichler P, Staber PB, Trneny M, Duell J, Waldron-Lynch M, Wagner S, Mukhopadhyay A, Dirnberger-Hertweck M, Burke JM, Nowakowski GS. Safety and efficacy of tafasitamab with or without lenalidomide added to first-line R-CHOP for DLBCL: the phase 1b First-MIND study. Blood. 2023 Oct 19;142(16):1348-1358. doi: 10.1182/blood.2023020637. PMID 37369099

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 33 | 33
Completed | 26 | 27
Not Completed | 7 | 6
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Progressive disease, joined another trial | 1 | 0
Not completed — Progressive disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.64) | 61.4 (12.34) | 62.6 (11.96)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 16 | 17 | 33
  65-84 years | 16 | 16 | 32
  Greater than or equal to 85 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 38
  Male | 15 | 13 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 33 | 64
  Other | 1 | 0 | 1
  Not Reported | 1 | 0 | 1
Weight at Baseline (kg) [Mean (Standard Deviation); unit: kg] | 73.03 (16.375) | 77.27 (16.016) | 75.15 (16.213)

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment-emergent Adverse Events (TEAEs)
Time Frame: 6 months approximately
Population: No participants in the "Arm A" Group were assessed for the "Patients with TEAE related to Lenalidomide only" row, since they did not receive Lenalidomide.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
Participants
  Patients with any TEAE | 33 | 33
  Patients with any study treatment-related TEAE | 31 | 32
  Patients with TEAE related to Tafasitamab only | 9 | 5
  Patients with TEAE related to Lenalidomide only: number analyzed (Participants) | 0 | 33
  Patients with TEAE related to Lenalidomide only |  | 16
  Patients with TEAE related to R-CHOP only | 29 | 23
  Patients with any grade ≥3 TEAE | 27 | 30
  Patients with any serious TEAE | 14 | 17

2. Secondary Outcome: Objective Response Rate (ORR) at the End of Treatment (EOT)
Description: The ORR at EOT was defined as the proportion of patients with Complete Response (CR) or Partial response (PR) based on the response achieved at the EOT Visit/early treatment discontinuation visit.
Time Frame: 6 months approximately
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
Participants | 25 | 27

3. Secondary Outcome: Metabolic, PET-negative Complete Response (CR) Rate at the End of Treatment
Time Frame: 6 months approximately
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
Participants | 24 | 22

4. Secondary Outcome: Incidence and Severity of Adverse Events (AEs) in the Follow-up (FU) Period
Time Frame: 18 months for non-treatment emergent adverse events, 6 months for treatment emergent adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
Participants
  Patients with at least 1 AE in the FU period | 26 | 26
  Patients with a Grade ≥3 TEAE in the FU period | 9 | 13
  Patients with at least 1 treatment related AE in the FU period | 9 | 7

5. Secondary Outcome: Best Objective Response Rate (ORR) Until the End of Study (EOS)
Description: The best ORR was defined as the proportion of patients with Complete Response (CR) or Partial Response (PR) as the best response until the EOS.
Time Frame: 24 months approximately
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
Participants | 30 | 31

6. Secondary Outcome: Metabolic, PET-negative Complete Response (CR) Rate Until the End of Study
Time Frame: 24 months approximately
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
Participants | 28 | 23

7. Secondary Outcome: Progression-free Survival (PFS) at 12 and 24 Months
Description: As many patients had their data censored, due to completing the study without disease progression or death due to any cause, the probability of PFS (%) was used.
Time Frame: 24 months approximately
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
percent
  Probability of PFS (%) at 12 months | 83.1 [64.0 to 92.6] | 76.8 [57.1 to 88.3]
  Probability of PFS (%) at 24 months | 72.7 [52.7 to 85.3] | 76.8 [57.1 to 88.3]

8. Secondary Outcome: Event-free Survival (EFS) at 12 and 24 Months
Description: As many patients had their data censored, due to completing the study without disease progression, death due to any cause, or the start of a new anti-lymphoma treatment, the probability of EFS (%) was used.
Time Frame: 24 months approximately
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
percent
  Probability of EFS (%) at 12 months | 77.4 [58.4 to 88.5] | 68.0 [48.6 to 81.4]
  Probability of EFS (%) at 24 months | 67.7 [48.4 to 81.2] | 68.0 [48.6 to 81.4]

9. Secondary Outcome: Time to Next Anti-lymphoma Treatment (TTNT)
Description: As many patients had their data censored, due to completing the study without needing to receive another anti-lymphoma treatment, the Probability of TTNT (%) was used. Time to next anti-lymphoma treatment survival % estimate was the estimated probability that a patient remained TTNT-free up to the specified point in time.
Time Frame: 24 months approximately
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
percent
  Probability of TTNT (%) at 12 months | 77.4 [58.4 to 88.5] | 71.9 [52.9 to 84.3]
  Probability of TTNT (%) at 24 months | 71.0 [51.6 to 83.7] | 68.8 [49.7 to 81.8]

10. Secondary Outcome: Overall Survival at 12 and 24 Months
Description: As many patients had their data censored, due to completing the study without death from any cause, the probability of OS (%) was used.
Time Frame: 24 months approximately
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 33 | 33
percent
  Probability of OS (%) at 12 months | 90.3 [72.9 to 96.8] | 93.8 [77.3 to 98.4]
  Probability of OS (%) at 24 months | 90.3 [72.9 to 96.8] | 93.8 [77.3 to 98.4]

11. Secondary Outcome: Anti-tafasitamab Antibodies Formation
Time Frame: 12 months approximately
Population: One patient in the Tafasitamab in addition to R-CHOP arm (Arm A) was missing a baseline sample and therefore could not be included in this analysis. In addition, no post-baseline evaluation was available for one patient in Arm A and one patient in Arm B hence the number of analyzed participants differs from overall.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 32 | 33
Participants
  Patients with pre-existing anti-tafasitamab antibodies | 1 | 0
  Patients without anti-tafasitamab antibodies after start of treatment: number analyzed (Participants) | 31 | 32
  Patients without anti-tafasitamab antibodies after start of treatment | 30 | 32
  Patients with anti-tafasitamab antibodies after the start of treatment: number analyzed (Participants) | 31 | 32
  Patients with anti-tafasitamab antibodies after the start of treatment | 1 | 0
  Patients with treatment-induced anti-tafasitamab antibodies: number analyzed (Participants) | 31 | 32
  Patients with treatment-induced anti-tafasitamab antibodies | 0 | 0
  Patients with treatment-boosted anti-tafasitamab antibodies: number analyzed (Participants) | 31 | 32
  Patients with treatment-boosted anti-tafasitamab antibodies | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months for non-treatment emergent adverse events, 6 months for treatment emergent adverse events, and approximately 24 months for all-cause mortality.
Description: Any AE reported from the treatment start date through 30 days after the last dose of treatment end date.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 4/33 | 2/33
Serious Adverse Events (participants affected / at risk) | 14/33 | 17/33
Other Adverse Events (participants affected / at risk) | 31/33 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=33) | Arm B (N=33)
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Generalized tonic-clonic seizure (Nervous system disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Device-related thrombosis (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Paraspinal abscess (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Infusion-related reaction (Injury, poisoning and procedural complications) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=33) | Arm B (N=33)
Neutropenia (Blood and lymphatic system disorders) | 18 | 26
Anaemia (Blood and lymphatic system disorders) | 16 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 14
Leukopenia (Blood and lymphatic system disorders) | 10 | 9
Lymphopenia (Blood and lymphatic system disorders) | 4 | 8
Stomatitis (Gastrointestinal disorders) | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 10 | 11
Nausea (Gastrointestinal disorders) | 10 | 9
Constipation (Gastrointestinal disorders) | 10 | 8
Vomiting (Gastrointestinal disorders) | 10 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Neuropathy peripheral (Nervous system disorders) | 9 | 10
Dysgeusia (Nervous system disorders) | 4 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 2
Paraesthesia (Nervous system disorders) | 1 | 2
Aphasia (Nervous system disorders) | 2 | 0
Asthenia (General disorders) | 6 | 8
Fatigue (General disorders) | 11 | 5
Oedema peripheral (General disorders) | 2 | 4
Oral candidiasis (Infections and infestations) | 2 | 2
Oral herpes (Infections and infestations) | 1 | 2
Infusion-related reaction (Injury, poisoning and procedural complications) | 7 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 9
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sinus tachycardia (Cardiac disorders) | 2 | 0
Weight decreased (Investigations) | 5 | 0
C-reactive protein increased (Investigations) | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5
Vertigo (Ear and labyrinth disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 9 | 6
Hypotension (Vascular disorders) | 5 | 5
Haemorrhoids (Gastrointestinal disorders) | 2 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 4
Dizziness (Nervous system disorders) | 2 | 3
Syncope (Nervous system disorders) | 2 | 0
Malaise (General disorders) | 0 | 3
Pyrexia (General disorders) | 5 | 2
Infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 2
Conjunctivitis (Infections and infestations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Folate deficiency (Metabolism and nutrition disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Hypertension (Vascular disorders) | 2 | 3
Weight increased (Investigations) | 2 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No investigator or institution may publish any results of the trial conducted at their site, before a first multicentre publication is made which covers the data from all sites. The author must coordinate the publication with the sponsor, who has the right to review it at least 60 days before their submission. If publication would affect the patentability of any invention to which the sponsor has rights, the sponsor can request to delay the proposed publication for no more than 90 days.

DOCUMENTS (2):
  • Study Protocol (2020-02-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT04134936/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT04134936/SAP_001.pdf